CLINICAL TRIAL: NCT05869669
Title: A Phase 2b Clinical Study of the P38 Alpha Kinase Inhibitor Neflamapimod in Patients With Dementia With Lewy Bodies
Brief Title: RewinD-LB - Clinical Study of Neflamapimod in Patients With Dementia With Lewy Bodies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Worldwide Clinical Trials (Other); CervoMed, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIP21-NFD-504; R01AG080536 (NIH); 2023-504373-20 (EudraCT Number)
Record Dates: First submitted 2023-04-12; First posted 2023-05-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Dementia With Lewy Bodies
Keywords: DLB
MeSH Terms: conditions — Lewy Body Disease | interventions — VX-745

STUDY DESIGN:
Intervention Model Description: Phase 2b (hypothesis-testing), multi-center, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neflamapimod (Active Comparator): Neflamapimod will be administered with food for 16 weeks in subjects with DLB. Subjects will receive 3 capsules per day (TID) with food (i.e., with the morning, mid-day and evening meals).
  Interventions: Drug: Neflamapimod
- Placebo (Placebo Comparator): Placebo will be administered with food for 16 weeks in subjects with DLB. Subjects will receive 3 capsules per day (TID) with food (i.e., with the morning, mid-day and evening meals).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neflamapimod — Neflamapimod is a highly specific inhibitor of the intra-cellular enzyme mitogen-activated protein kinase14 (p38α) provided in 40mg capsules
  Other Names: VX-745
  Arms: Neflamapimod
Drug: Placebo — Placebo is a capsule that looks just like neflamapimod but without the active ingredients
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether neflamapimod can improve learning skills, problem solving skills, and memory loss in people diagnosed with DLB. More specifically, improvement in verbal learning, memory, and attention, as well as cognitive and functional performance will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥55 years.
2. Subject or subject's legally authorized representative is willing and able to provide written informed consent.
3. 3. Probable DLB by consensus criteria (McKeith et al, 2017), including a positive DaTscan™. Specifically, the subject must have the presence of dementia in association with:

   * At least two (2) core clinical features (fluctuating cognition, visual hallucinations, REM sleep disorder, and/or parkinsonism); or
   * One (1) core clinical feature plus an abnormal DaTscan™. Historical polysomnography (PSG)-verified REM sleep behavioral disorder (RBD), FDG-PET imaging, or MIBG myocardial scintigraphy can take the place of an abnormal DaTscan™ in a patient with only one core clinical feature.
4. CDR Global Score 0.5 (very mild dementia) or 1.0 (mild dementia) during Screening
5. Background dementia therapy:

   * Not currently receiving cholinesterase inhibitor therapy. If the patient received such therapy previously, that therapy must have been discontinued at least 3 months prior to randomization.
   * Receiving cholinesterase inhibitor therapy alone. If the patient is currently receiving cholinesterase inhibitor therapy, the patient must have received such therapy for greater than 3 months and on a stable dose for at least 6 weeks at the time of randomization. Except for reducing the dose for tolerability reasons, the dose of cholinesterase inhibitor may not be modified during the study.
   * Memantine therapy is allowed, if it had been started at least 3 months prior to randomization and the patient is also receiving cholinesterase inhibitor therapy. If the patient has never been on cholinesterase inhibitor therapy (naïve), then memantine monotherapy is allowed.
6. Normal or corrected eyesight and auditory abilities, sufficient to perform all aspects of the cognitive and functional assessments.
7. No history of learning difficulties that may interfere with their ability to complete the cognitive tests.
8. Received vaccination for SARS-CoV-19 unless medical contraindications prevent being vaccinated, or has a history of natural infection.
9. Must have reliable informant or caregiver.

Exclusion Criteria:

1. Diagnosis of any other ongoing central nervous system (CNS) condition other than DLB, including, but not limited to, post-stroke dementia, vascular dementia, Alzheimer's disease (AD), or Parkinson's disease (PD).
2. Plasma ptau181 result above the threshold that indicates evidence of pathology associated with Alzheimer's disease at Screening.
3. Suicidality, defined as active suicidal thoughts within 6 months before Screening or at Baseline, defined as answering yes to items 4 or 5 on the C-SSRS, or history of suicide attempt in previous 2 years, or, in the Investigator's opinion, at serious risk of suicide.
4. Ongoing major and active psychiatric disorder and/or other concurrent medical condition that, in the opinion of the Investigator, might compromise safety and/or compliance with study requirements.
5. Diagnosis of alcohol or drug abuse within the previous 2 years.
6. Poorly controlled clinically significant medical illness, such as hypertension (blood pressure >180 mmHg systolic or 100 mmHg diastolic); myocardial infarction within 6 months; uncompensated congestive heart failure or other significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would interfere with assessment of drug safety.
7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 × the upper limit of normal (ULN), total bilirubin >1.5 × ULN, and/or International Normalized Ratio (INR) >1.5. If patient is taking blood thinners (e.g., warfarin), and has no known liver issues, INR >3.
8. Known human immunodeficiency virus, hepatitis B, or active hepatitis C virus infection.
9. Participated in a study of an investigational drug less than six weeks or 5 half-lives of an investigational drug, whichever is longer, before enrollment in this study.
10. History of previous neurosurgery to the brain within the past five years.
11. If male with female partner(s) of child-bearing potential, unwilling or unable to adhere to contraception requirements specified in the protocol.
12. If female who has not has not reached menopause >1 year previously or has not had a hysterectomy or bilateral oophorectomy/salpingo-oophorectomy, has a positive pregnancy test result during Screening and/or is unwilling or unable to adhere to the contraception requirements specified in the protocol.
13. Weight less than 50kg.

All participants who complete the initial 16-week period of the study will be able to continue in the study and receive neflamapimod for an additional 32 weeks (8 months) regardless of whether they received neflamapimod of placebo during the the first 16 weeks.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) in neflamapimod-treated subjects compared to placebo recipients. | 16 weeks
  The primary objective is to demonstrate the efficacy of neflamapimod, compared to placebo, as a treatment for DLB, as assessed by the CDR-SB scale.
  CDR-SB scores range from 0 to 18 with a higher score indicating worsening of cognitive impairment.

SECONDARY OUTCOMES:
Change in Timed Up and Go Test (TUG) in neflamapimod-treated subjects compared to placebo recipients. | 16 weeks
  Demonstrate that neflamapimod improves motor function in patients with DLB, compared to placebo, as assessed by the TUG test.
  TUG scores typically range from 6 to 20 seconds with a higher score indicating worse mobility. A score of >15 indicates an increased risk of falls.
Change in the composite score of the Neuropsychological Test Battery (NTB), including tests of attention, executive function, and visual learning in neflamapimod-treated subjects compared to placebo recipients. | 16 weeks
  Demonstrate that neflamapimod improves cognition, compared to placebo, as assessed by a DLB-specific NTB in patients with DLB. NTB includes Cogstate Detection test (DET), Cogstate Identification test (IDN), Cogstate One Card Learning test (OCL), Cogstate One Back test (ONB).
  Each score on the individual tests is converted to a z-score, and then a total z-score for the composite is calculated, in which each test is weighted equally. As the analysis is based on z-scores, there is no minimum or maximum value. A z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A positive change in z-score indicates an improvement in cognition and a negative change in z-score indicates a worsening in cognition.
Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-GCIC) score at Week 16 in neflamapimod-treated subjects compared to placebo recipients. | 16 weeks
  Demonstrate that neflamapimod improves global (cognition, function and behavior) disease status evaluated by a clinician with caregiver input, compared to placebo, in patients with DLB, as assessed ADCS-CGIC score.
  ADCS-CGIC scores range from 1 to 7, where 1 = marked improvement, 2= moderate improvement, 3 = minimal improvement, 4 = no change, 5 = minimal worsening, 6 = moderate worsening, and 7 = marked worsening.

OTHER OUTCOMES:
Exploratory outcome - Dementia Cognitive Fluctuations Scale (DCFS) | 16 weeks
  Change in DCFS score in neflamapimod-treated subjects compared to placebo recipients.
  DCFS scores range from 4 to 20 where a higher score indicates more severe cognitive fluctuations and disease worsening.
Exploratory outcome - 12-item Neuropsychiatric Inventory (NPI-12) | 16 weeks
  Change in neflamapimod-treated subjects compared to placebo recipients in the following:
  * Select domains of the NPI-12, including depression (dysphoria), apathy, hallucinations, and agitation/aggression.
  * Change in hallucinations frequency x severity score within the NPI-12 in subjects who report hallucinations at baseline.
  * Change in sleep and night-time behavior change within the NPI-12.
  NPI-12 scores range from 0 to 12 for each individual domain and 0 to 144 total score, where a higher score indicates worsening of neuropsychiatric symptoms.
Exploratory outcome - Movement Disorder Society - Unified Parkinson's Disease Rating Scale - Part III (MSD-UPDRS3) motor examination (Part III) | 16 weeks
  Change in MDS-UPDRS3 score in neflamapimod-treated subjects compared to placebo recipients..
  MDS-UPDRS 3 scores range from 0 to 108 where a higher score indicates more severe motor symptoms.
Exploratory outcome - EEG | 16 weeks
  Change in beta functional connectivity and in alpha reactivity on quantitative EEG in neflamapimod-treated subjects compared to placebo recipients..
  Functional connectivity will be analyzed as Amplitude Envelope Correlation (AECc), a measure of interregional communication within the brain. AECcs are computed by correlating the amplitude (energy) envelopes of oscillatory brain signals in two different brain regions. AECc ranges between 0 and 1, with higher AECc values indicating increased functional connectivity. In this study, the primary EEG evaluation will be AECc within the beta band (13-30 Hz), i.e. beta functional connectivity.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (29):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Banner Alzheimer's Institute - Edson Family Lewy Body Dementia Center, Tucson, Arizona
  - UCSD Health Sciences - Movement Disorders Center, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - SC3 Research Group, Pasadena, California
  - University of Colorado - Dept of Neurology, Aurora, Colorado
  - Georgetown Univ Hospital - Dept of Neurology, Washington D.C., District of Columbia
  - JEM Research Institute, Lake Worth, Florida
  - ClinCloud, Melbourne, Florida
  - AdventHealth Neuroscience Research, Orlando, Florida
  - Panhandle Research and Medical Clinic, Pensacola, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - Johns Hopkins School of Medicine - Dept of Neurology, Baltimore, Maryland
  - Mass General Hospital/Harvard Medical School - Dept of Neurology, Charlestown, Massachusetts
  - Mayo Clinic - Alzheimer's Disease Research Center, Rochester, Minnesota
  - University of Nebraska Medical Center - Dept of Neurological Sciences, Omaha, Nebraska
  - Cleveland Clinic - Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Columbia University - Taub Institute/Neurology Dept, New York, New York
  - University of North Carolina - Dept of Neurology, Chapel Hill, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - Cleveland Clinic - Center for Brain Health, Cleveland, Ohio
  - Ohio State University - Dept of Neurology, Columbus, Ohio
  - Center for Cognitive Health, Portland, Oregon
  - Houston Methodist Hospital - Stanley Appel Neurology Dept, Houston, Texas
  - Sana Research, Arlington, Virginia
  - Virginia Commonwealth University - Parkinson's and Movement Disorders Center, Richmond, Virginia
- Netherlands (3):
  - Brain Research Center - Den Bosch, 's-Hertogenbosch
  - Brain Research Center - Amsterdam, Amsterdam
  - Brain Research Center - Zwolle, Zwolle
- United Kingdom (8):
  - Belfast Health & Social Care Trust, Belfast
  - Cambridgeshire and Peterborough NHS Foundation Trust, Fulbourn Hospital - Windsor Research Unit, Cambridge
  - South London and Maudsley NHS Foundation Trust, London
  - Re:Cognition Health, London
  - University College London (UCL) Clinical Research Facility, University College London Hospitals NHS Foundation Trust, London
  - Campus Ageing Research Unit (CARU) - Newcastle upon Tyne, CNTW NHS Foundation Trust, Newcastle upon Tyne
  - Cornwall Partnership NHS Foundation Trust (University of Exeter), Redruth
  - Memory Assessment and Research Centre (MARC) - Moorgreen Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol: EIP21-NFD-504 Ex-US Protocol version (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT05869669/Prot_000.pdf
  • Study Protocol: EIP21-NFD-504 US Protocol version (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT05869669/Prot_001.pdf
  • Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT05869669/SAP_002.pdf